CLINICAL TRIAL: NCT07299357
Title: Prospective Observational Trial of Image-guided Ablative STereotactic bOdy Radiation Therapy for Primary kidNey Cancer: the STONE Trial
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: STONE TRIAL
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Renal Cancer
Keywords: renal cancer; stereotactic body radiotherapy; radiotherapy; cancer treatment; renal cancer treatment; surgery
MeSH Terms: conditions — Kidney Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT) — high dose radiation in few fractions

SUMMARY:
The study objective is to evaluate the use of Stereotactic Body Radiotherapy (high dose of radiation in a few fractions) to cure primary renal cancer in those patients that are not indicated to surgery (high risk of complications, refusal of the patient). This therapy is already used in clinical setting for many tumors with good tolerance as it is not invasive, does not require anesthesia and hospitalization making it suitable for elderly people and frail patients. However there are not enough information regarding the use of ablative doses for the cure of renal cancer and for this reason this study aims to support the use of Stereotactic Body Radiotherapy as a standard of care for inoperable primary renal tumor. This is an observational study, so it collects data from clinical pratice only and does not request study specific procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ECOG performance status 0 - 2
* Histologically confirmed diagnosis of primary RCC
* cT1 stage tumor with single lesion with maximum diameter of 7 cm
* Medically inoperable or at high risk of complication from surgery, or declined surgery
* Absence of metastatic disease
* Written informed consent

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) < 30 mls/min
* Previous radiotherapy on the same site
* Previous systemic therapy for RCC
* Tumor diameter larger than 7 cm
* Presence of metastatic disease
* Life expectancy < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with renal cancer not candidate to surgery
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
evaluate LC of treated lesions at 1 year | from end of treatment to 1 year
  local progression is defined as an enlargement of at least 20% relative and 5 mm absolute increase of sum of diameters of target lesions compared to baseline at least after 6 months from treatment end

SECONDARY OUTCOMES:
to assess acute and late toxicity | from start of treatment to 3 years
  evaluate the presence of toxicities to treatment according to CTCAE 4.03
To assess kidney function with serum creatinine | from start of treatment to 3 years
  evaluating serum creatinine at each follow up visit through blood analysis (mg/dL)
Progression Free Survival (PFS) | from end of treatment to 1 year
  to asses through standard imaging according to clinical practice - The length of time during and after the treatment of cancer that a patient lives with the disease but it does not get worse
metastasis free survival | from end of treatment to 3 years
  to asses through standard imaging according to clinical practice - The length of time from the start of treatment for cancer that a patient is still alive and the cancer has not spread to other parts of the body
Overall Survival | from end of treatment to 3 years
  to asses through standard imaging according to clinical practice - The length of time from the start of cancer treatment during which patients diagnosed with the disease are still alive.
To asses Quality of Life | from start of treatment to 3 years
  Through QLQ-C30 questionnarie we will evaluate quality of life, patient will answer different questions crossing the number that is more suitable regarding their condition (the patient can respond by crossing a number from 1 to 4, 1 = excellent quality of life, 4 = terrible quality of life)
To assess kidney function with estimated glomerular filtration rate | from start of treatment to 3 years
  evaluating eGFR at each follow up visit through blood analysis (ml/min)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Humanitas PIO X, Milan, Milan
  - Irccs Humanitas Research Hospital, Rozzano, Milan

REFERENCES:
- [Background] Siva S, Bressel M, Sidhom M, Sridharan S, Vanneste BGL, Davey R, Montgomery R, Ruben J, Foroudi F, Higgs B, Lin C, Raman A, Hardcastle N, Hofman MS, De Abreu Lourenco R, Shaw M, Mancuso P, Moon D, Wong LM, Lawrentschuk N, Wood S, Brook NR, Kron T, Martin J, Pryor D; FASTRACK II Investigator Group. Stereotactic ablative body radiotherapy for primary kidney cancer (TROG 15.03 FASTRACK II): a non-randomised phase 2 trial. Lancet Oncol. 2024 Mar;25(3):308-316. doi: 10.1016/S1470-2045(24)00020-2. PMID 38423047
- [Background] Siva S, Ali M, Correa RJM, Muacevic A, Ponsky L, Ellis RJ, Lo SS, Onishi H, Swaminath A, McLaughlin M, Morgan SC, Cury FL, Teh BS, Mahadevan A, Kaplan ID, Chu W, Grubb W, Hannan R, Staehler M, Warner A, Louie AV. 5-year outcomes after stereotactic ablative body radiotherapy for primary renal cell carcinoma: an individual patient data meta-analysis from IROCK (the International Radiosurgery Consortium of the Kidney). Lancet Oncol. 2022 Dec;23(12):1508-1516. doi: 10.1016/S1470-2045(22)00656-8. Epub 2022 Nov 16. PMID 36400098
- [Background] AIOM-AIRTUM. I numeri del cancro in Italia. Rapporto 2020. Disponibile sul sito: https://www.aiom.it/i-numeri-del-cancro-in-italia